CLINICAL TRIAL: NCT04350372
Title: The MitraClip Russia Trial: A Prospective, Single-Center, Single-Arm Clinical Evaluation of the MitraClip System for the Treatment of Mitral Regurgitation
Brief Title: MitraClip Russia Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABT-CIP 10334
Record Dates: First submitted 2020-04-08; First posted 2020-04-17 (Actual); Results first posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Functional Mitral Regurgitation; Degenerrative Mitral Regurgitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- MitraClip (Experimental): Subject will receive MitraClip procedure with MitraClip NT System
  Interventions: Device: MitraClip Procedure

INTERVENTIONS:
Device: MitraClip Procedure — MitraClip procedure with MitraClip NT System

SUMMARY:
The MitraClip System is the first commercially available catheter-based option for the treatment of MR. The MitraClip System was developed as an alternate percutaneous technology which may serve as a viable therapeutic option for patients at high risk for open-heart surgery. Treatment with the MitraClip device allows patients to undergo a less invasive procedure that can mechanistically reduce MR and allow for improved quality of life. The MitraClip procedure is performed under general anesthesia without the use of a heart-lung machine, with recovery typically lasting two to three days.

The objective of this study is to evaluate safety and effectiveness of the MitraClip NT procedure in the Russian population for treatment of Mitral Regurgitation.

DETAILED DESCRIPTION:
Mitral regurgitation (MR) is the most common heart valve condition in the world. MR occurs when the mitral valve does not close properly, allowing blood to leak back into the upper chamber of the heart. As a result, the heart may try to pump harder in order to compensate for the decrease in blood flow to the rest of the body. Patients with severe MR suffer from debilitating symptoms such as shortness of breath, heart palpitations, lightheadedness, and fatigue. These patients are at risk of poor quality of life, marked limitation in activity, repeated heart failure hospitalizations, and increased mortality. Chronic severe MR is often associated with heart failure and can lead to death if left untreated.

While mitral valve repair or replacement surgery is currently regarded as standard of care, many patients with clinically significant MR are at an unacceptable risk of morbidity and mortality and are therefore not appropriate surgical candidates. To optimize afterload reduction and treatment of fluid load, these patients are often treated with medical management (i.e., beta blockers, ACE inhibitors, angiotensin II receptor blockers) which may relieve MR symptoms, but does not address the underlying cause of the condition. As a result, a significant portion of patients treated medically continue to progress to heart failure and experience an increasingly debilitating quality of life. A significant unmet clinical need thus exists for the treatment of moderate-to-severe and severe MR in high surgical risk patients.

The MitraClip System has been in clinical use for treatment of significant MR since 2003. The device received CE (Conformité Européenne) Mark for both DMR and FMR indications in March 2008 and was approved by FDA for DMR indication in October 2013 and for FMR indication in March 2019. The system is approved for use in more than 80 countries or regions. More than 80,000 patients have undergone the MitraClip procedure worldwide, with the majority of experience in high surgical risk patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Symptomatic moderate-to-severe (3+) or severe MR (4+) chronic DMR or FMR determined by assessment of a qualifying transthoracic echocardiogram (TTE) obtained within 90 days or transesophageal echocardiogram (TEE) obtained within 180 days prior to subject registration.
* LVEF ≥ 30%
* NYHA classification is class II, class III, or ambulatory class IV.
* Subject is deemed difficult for mitral valve surgery due to either STS surgical mortality risk for mitral valve replacement of ≥ 8% OR due to the presence of one of the following risk factors (Porcelain aorta or mobile ascending aortic atheroma, Post-radiation mediastinum, Previous mediastinitis, Functional MR with LVEF<40%, Over 75 years old with LVEF<40%, Re-operation with patent grafts, Two or more prior cardiothoracic surgeries, Hepatic cirrhosis, Other surgical risk factor(s))
* Mitral valve area ≥ 4.0 cm2.
* The primary regurgitant jet is non-commisural, and in the opinion of the implanting investigator can successfully be treated by the MitraClip NT System. If a secondary jet exists, it must be considered clinically insignificant

Exclusion Criteria:

* Subject is currently participating in another clinical investigation
* Pregnant or nursing subjects and those who plan pregnancy during the clinical investigation follow up period
* Patients with the following conditions: Patients who cannot tolerate procedural anticoagulation or post procedural anti-platelet regimen; Active endocarditis of the mitral valve; Rheumatic mitral valve disease; Evidence of intracardiac, inferior vena cava (IVC) or femoral venous thrombus.
* Contraindications for reusable accessories (stabilizer, lift, support plate)
* Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness of the clinical investigation results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2020-09-24 (Actual); Study Completion 2020-10-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- FSBI "NICC of Cardiology" of the Ministry, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MitraClip
Started | 16
Completed | 15
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | MitraClip
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.1 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Russia | 16
Height [Mean (Standard Deviation); unit: cm] | 168.7 (11.9)
Weight [Mean (Standard Deviation); unit: Kg] | 81.3 (21.1)
Patients with Society of Thoracic Surgeons (STS) Mitral Valve Replacement Score >= 8% [Count of Participants; unit: Participants] — The STS MV Replacement score is a validated risk-prediction model for MV Replacement on data from the STS National Adult Cardiac Surgery Database.
  As of November 15, 2018, The Society of Thoracic Surgeons released an updated short-termrisk calculator to reflect the latest 2018 adult cardiac surgery risk models. The STS Calculator allows you to calculate a patient's risk of Mitral Valve Replacement for the most commonly performed cardiac surgeries.
  Participants | 7
Mitral Regurgitation [Count of Participants; unit: Participants]
  3+ (Moderately Severe) | 7
  4+ (Severe) | 9
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 28.19 (4.28)
Society of Thoracic Surgeons (STS) Mitral Valve [Mean (Standard Deviation); unit: Percentage of Risk] — The STS score is a validated risk-prediction model for open surgerybased on data from the STS National Adult Cardiac Surgery Database. In general, an STSpredicted risk of surgical mortality of 4%-8% is considered intermediate risk and 8% orgreater is considered high risk.
  As of November 15, 2018, The Society of Thoracic Surgeons released an updated short-termrisk calculator to reflect the latest 2018 adult cardiac surgery risk models. The STS Calculator allows you to calculate a patient's risk of mortality and morbidities for the most commonlyperformed cardiac surgeries.
  Percentage of Risk | 6.33 (3.94)
BNP [Mean (Standard Deviation); unit: pg/mL] — Population: All the available data have been reported.
  pg/mL
    number analyzed (Participants) | 10
    (all) | 532.71 (562.18)
NT proBNP [Mean (Standard Deviation); unit: pg/mL] — Population: All the available data have been reported.
  pg/mL
    number analyzed (Participants) | 15
    (all) | 2426.87 (2706.58)
Serum Creatinine [Mean (Standard Deviation); unit: mg/dL] | 1.34 (0.40)
Effective Regurgitant Orifice Area (EROA) [Mean (Standard Deviation); unit: cm^2] | 0.39 (0.14)
Regurgitant Volume (RV) [Mean (Standard Deviation); unit: mL/beat] | 53.6 (9.0)
Regurgitant Fraction (RF) [Mean (Standard Deviation); unit: %] — Population: All the available data have been reported.
  %
    number analyzed (Participants) | 15
    (all) | 58.9 (16.4)
Mitral Valve Area (MVA) [Mean (Standard Deviation); unit: cm^2] | 5.53 (0.57)
Left Ventricular Ejection Fraction (LVEF) [Mean (Standard Deviation); unit: %] | 46.1 (12.0)
Left Ventricular End Systolic Dimension (LVESD) [Mean (Standard Deviation); unit: cm] | 4.47 (0.91)
Ventricular End Diastolic Dimension (LVEDD) [Mean (Standard Deviation); unit: cm] | 6.05 (0.77)
Left Ventricular End Systolic Volume (LVESV) [Mean (Standard Deviation); unit: mL] | 93.8 (49.0)
Left Ventricular End Diastolic Volume (LVEDV) [Mean (Standard Deviation); unit: mL] | 158.9 (46.3)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Successful Implantation of the MitraClip NT Device
Description: Successful implantation of the MitraClip NT device resulting in a decrease in the MR severity grade as assessed from the discharge echocardiogram (10-day echocardiogram will be used if discharge is unavailable or uninterpretable). Subjects who die or undergo mitral valve surgery before discharge will be considered a failure for the procedure
Time Frame: 30-day
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip
Number analyzed (Participants) | 16
Participants | 15

ADVERSE EVENTS:
Time Frame: 30 Days
Arm/Group | MitraClip
All-Cause Mortality (participants affected / at risk) | 1/16
Serious Adverse Events (participants affected / at risk) | 2/16
Other Adverse Events (participants affected / at risk) | 2/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MitraClip (N=16)
Iatrogenic ASD with Complications (General disorders) | 1 (1)
Stroke (General disorders) | 1 (1)
Cardiac arrest takotsubo cardiomyopathy (General disorders) | 1 (1)
Pneumonia (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MitraClip (N=16)
Single Leaflet Device Attachment (SLDA) (General disorders) | 1 (1)
furuncle on chest (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-11-15): https://cdn.clinicaltrials.gov/large-docs/72/NCT04350372/Prot_002.pdf
  • Statistical Analysis Plan (2021-11-19): https://cdn.clinicaltrials.gov/large-docs/72/NCT04350372/SAP_003.pdf